CLINICAL TRIAL: NCT00948155
Title: Assessment of Smoking Topography and Behaviors During Response to Varenicline
Brief Title: Measuring Smoking Behaviors While Using Varenicline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Andrew Strasser, Associate Professor Department of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 808930
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Nicotine Dependence
Keywords: smoking; nicotine; varenicline
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline before placebo (Experimental): Drug (Varenicline (Chantix)): Placebo
  Intervention to be administered is: participants will receive standard dosing regimen of Varenicline for 21 days total, followed by 14-day washout and 21 days of placebo. Standard dosing: 0.5 mg days 1-3; 0.5 mg bid days 4-7; 1.0 mg bid days 8-21.
  Interventions: Drug: Varenicline
- Placebo then Varenicline (Experimental): Placebo: Drug Varenicline (Chantix)
  Intervention to be administered is: participants will receive 21 days of placebo, followed by 14-day washout and standard dosing regimen of Varenicline for 21 days total. Standard dosing: 0.5 mg days 1-3; 0.5 mg bid days 4-7; 1.0 mg bid days 8-21.
  Intervention 'Drug (Varenicline (Chantix)): Placebo'
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Intervention Drug (Varenicline (Chantix) will be administered in standard dosing in pill format: 0.5 mg days 1-3; 0.5 mg bid daily days 4-7; 1.0 mg bid daily days 8-21.
  Other Names: Chantix

SUMMARY:
This study will demonstrate the behavioral responses to varenicline, helping to better understand its mechanisms. Hypotheses for the study are to observe decreases in smoking topography and nicotine cigarette choice on varenicline, relative to placebo; and decreases on day 21 relative to day 7 during varenicline treatment. We also propose to examine if extended duration of treatment has clinical significance in decreasing smoking behaviors, thus increasing the efficacy of varenicline.

DETAILED DESCRIPTION:
This study is designed to examine the behavioral responses a cigarette smoker may have to using varenicline. Behavioral responses may help to better understand its mechanisms which in turn could improve treatment outcomes. The primary hypothesis for the study is to observe decreases in smoking topography, an objective measure of smoking behavior or puffing, on varenicline, relative to placebo; and decreases on day 21 relative to day 7 during varenicline treatment. We will also examine puffing and nicotine cigarette choices during lab visits at baseline, and Days 7 and 21. We also propose to examine if extended duration of treatment has clinical significance in decreasing smoking behaviors, thus potentially increasing the efficacy of varenicline.

ELIGIBILITY:
Inclusion Criteria:

* self report minimum 10 daily cigarettes
* self report smoking every day past 5 years
* between the ages 21-65
* self report intention to try to quit smoking in the next 6 months

Exclusion Criteria:

* self reported use of any nicotine-containing products other than non-menthol cigarettes
* self reported history or current treatment of substance abuse (other than nicotine dependence)
* self reported alcohol use greater than 25 standard drinks per week;
* currently pregnant, planned pregnancy or lactating (females: negative urine pregnancy screen)
* self reported history or current diagnosis of any Axis 1 disorders except past depression
* self reported serious or unstable disease within past year
* self reported history of epilepsy or seizure disorder;
* self reported history or current diagnosis of COPD (chronic obstructive pulmonary disease), cardiovascular disease, heart attack, or uncontrolled hypertension
* self reported kidney function impairment
* any current or recent (30 day) use of: smoking cessation medications, anti-psychotics, anti-depressants, anti-anxiety, panic medications, stimulants or opiate-containing medications
* less than 5 years of daily smoking
* any medical condition or concomitant medication that could compromise participant safety or treatment
* provide a baseline carbon monoxide (CO) reading < 10 ppm
* self reported use of non filtered cigarettes
* inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Tobacco Use Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Ashare RL, Tang KZ, Mesaros AC, Blair IA, Leone F, Strasser AA. Effects of 21 days of varenicline versus placebo on smoking behaviors and urges among non-treatment seeking smokers. J Psychopharmacol. 2012 Oct;26(10):1383-90. doi: 10.1177/0269881112449397. Epub 2012 Jun 13. PMID 22695488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in a research laboratory in a school of medicine. Dates of recruitment: first participant first visit March 31, 2009; last participants last visit December 02, 2010
Pre-assignment Details: 48 participants signed consents and were enrolled in the study. Medical clearance was achieved by 41; 29 returned for the first laboratory visit which is the first day drug/placebo was administered. The 12 who did not return for the Day 1 visit were not included further in the study.
  There was a minimum 14 washout period between drug conditions.
Groups:
- Placebo Then Varenicline: Participants will receive 21 days of placebo, followed by 14-day washout and standard dosing regimen of Varenicline for 21 days total. Standard dosing: 0.5 mg days 1-3; 0.5 mg bid days 4-7; 1.0 mg bid days 8-21.
  Varenicline (Chantix) : Standard dosing in pill format: 0.5 mg days 1-3; 0.5 mg bid daily days 4-7; 1.0 mg bid daily days 8-21.
- Varenicline Before Placebo: Participants will receive standard dosing regimen of Varenicline for 21 days total, followed by 14-day washout and 21 days of placebo. Standard dosing: 0.5 mg days 1-3; 0.5 mg bid days 4-7; 1.0 mg bid days 8-21.
  Varenicline (Chantix) : Standard dosing in pill format: 0.5 mg days 1-3; 0.5 mg bid daily days 4-7; 1.0 mg bid daily days 8-21.
Period: First Intervention 21 Days
Arm/Group | Placebo Then Varenicline | Varenicline Before Placebo
Started | 14 | 15
Completed | 12 | 13
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: Washout 14 Days
Arm/Group | Placebo Then Varenicline | Varenicline Before Placebo
Started | 12 | 13
Completed | 11 | 11
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Period: Second Intervention 21 Days
Arm/Group | Placebo Then Varenicline | Varenicline Before Placebo
Started | 11 | 11
Completed | 9 | 8
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Varenicline | Varenicline Before Placebo | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.7) | 37.6 (12.8) | 39.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Smoking Topography: Total Puff Volume
Description: Total puff volume was created by summing all of the puffs from the cigarette smoked in the lab at each time point (each lab visit). This value represents the total volume of smoke extracted from a single cigarette and it a standard measure of smoking behavior. A total puff volume represents the total smoking volume from a cigarette. Values are reported in milliliters. Value of interest is the average puff volume across all sessions for all participants in a group and is reported as a key measure of smoking behavior. Analyses were repeated measures analysis of variance where individual, time and drug were within factors.
Time Frame: Days 1-21 of each of 2 study periods
Population: All those participants who completed both study periods were included in the analysis.
Measure: Mean (Standard Error); unit: milliliters
Arm/Group | Placebo Then Varenicline | Varenicline Before Placebo
Number analyzed (Participants) | 9 | 8
milliliters | 523.4 (41) | 684.6 (33)

2. Primary Outcome: The Number of Choices of a Nicotine Containing Cigarette Compared to a Non-nicotine Cigarette.
Description: Participants were given 4 puff choices (between a nicotine containing and de-nicotinized cigarette) on 6 study visits, for a total of 24 choices. Number of puffs reported is average across both study periods.
Time Frame: Days 1, 7, 21 of each of two 21 day study periods
Population: All participants who completed the task were included in the analysis
Measure: Mean (Standard Error); unit: number of puffs chosen of a maximum 24
Arm/Group | Placebo Then Varenicline | Varenicline Before Placebo
Number analyzed (Participants) | 9 | 8
number of puffs chosen of a maximum 24 | 12 (4.5) | 11.5 (5.1)

3. Primary Outcome: Daily Cigarette Consumption
Description: Average of the number of cigarettes smoked per day
Time Frame: Two 21 day study periods
Measure: Mean (Standard Error); unit: number of cigarettes smoked per day
Groups:
- Placebo: 21 days using placebo
- Varenicline: 21 days using Varenicline
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 17
number of cigarettes smoked per day
  Start of 21 day period | 16.2 (1.4) | 16.1 (0.86)
  End of 21 day period | 14.4 (1.2) | 12.8 (1.3)

4. Secondary Outcome: Total Nicotine Metabolites From Urine Samples
Description: Total urinary metabolites from urine samples collected at Day 1 and Day 21
Time Frame: Samples from Day 1 and Day 21 of two 21 day Periods
Population: Subjects who completed both 21 day placebo and drug periods.
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 17
micromolar
  Day 1 | 110 (14) | 111 (15)
  Day 21 | 79 (14) | 81 (9)

5. Secondary Outcome: Nicotine Levels From Urine Samples
Description: Nicotine levels from urine samples collected at Day 1 and Day 21.
Time Frame: Samples from Day 1 and Day 21 of two 21 day Periods
Population: Subjects who completed both 21 day placebo and drug periods.
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 17
micromolar
  Day 1 | 20.0 (6) | 24.0 (5)
  Day 21 | 18.0 (6) | 13.8 (3)

6. Secondary Outcome: Cotinine Levels From Urine Samples
Description: Cotinine levels from urine samples collected at Day 1 and Day 21.
Time Frame: Samples from Day 1 and Day 21 of two 21 day Periods
Population: Subjects who completed both 21 day placebo and drug periods.
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 17
micromolar
  Day 1 | 19.0 (2) | 16.9 (2)
  Day 21 | 12.0 (2) | 14.0 (2)

7. Secondary Outcome: Carbon Monoxide Levels
Description: Exhaled breath carbon monoxide levels collected at Day 1 and Day 21 sessions. Alveolar carbon monoxide is a validated assessment of smoke exposure.
Time Frame: Samples from Day 1 and Day 21 of two 21 day Periods
Population: Subjects who completed both 21 day placebo and drug periods.
Measure: Mean (Standard Error); unit: parts per million
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 17
parts per million
  Day 1 | 30 (4) | 23.2 (2)
  Day 21 | 25 (2) | 22 (2)

8. Secondary Outcome: Subjective Measures to Assess Smoking Urges
Description: Craving for cigarettes was assessed with the 32-item Questionnaire of Smoking Urges (QSU) during each study visit. In order to calculate the QSU measure, each item is rated on a Likert-type scale from 1 (strongly disagree) to 7 (strongly agree). The values are then summed to create a single total score. Well validated 2 factor subscale scores were also created by summing the item scores for the 2 factors: Factor 1 reflects the desire to smoke for pleasure and Factor 2 reflects urges to smoke to relieve withdrawal-related negative affect. Internal consistency for each scale across all time points was high (Cronbach's α > 0.95, 0.85, and 0.95 for Factor 1, Factor 2, and QSU total, respectively). Scale range is 1-7 where 1 is low urge to smoke and 7 represents high urge to smoke. Data was collected at each time point but outcome measure of interest is end of period.
Time Frame: Days 21 of each of the two 21-day study periods, range 1(low)-7(high)
Population: Subjects who completed both 21 day placebo and drug periods.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 17
units on a scale
  Factor 1 Day 1 | 4.2 (0.7) | 4.3 (0.6)
  Factor 1 Day 21 | 3.9 (0.6) | 3.7 (0.4)
  Factor 2 Day 1 | 2.5 (0.3) | 2.8 (0.3)
  Factor 2 Day 21 | 2.4 (0.4) | 2.6 (0.3)

ADVERSE EVENTS:
Description: Systematic assessment of adverse events occurred at baseline, Days 1, 7, 21 when participant is present in research center.
Arm/Group | Placebo Then Varenicline | Varenicline Before Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

LIMITATIONS AND CAVEATS:
Attrition rates were high. The final sample consisted primarily of Caucasian males, which may limit the generalizability of the present findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No